CLINICAL TRIAL: NCT06491576
Title: A Single-center, Randomized, Double-blind, Multiple Ascending Dose, Placebo-controlled Phase Ib/IIa Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Early Pharmacodynamics of BGT-002 Tablets in Subjects With NASH
Brief Title: A Clinical Trial of BGT-002 Tablets in Subjects With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Burgeon Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGT-002-004
Record Dates: First submitted 2024-05-30; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: NASH

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental)
  Interventions: Drug: BGT-002
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGT-002 — taking the study drug orally
  Arms: Test Group
Drug: Placebo — taking the placebo orally
  Arms: Placebo Group

SUMMARY:
This study is a single-center, randomized, double-blind, multiple ascending doses (MAD), placebo-controlled phase Ib/IIa clinical trial of BGT-002 Tablets in subjects with NASH to evaluate the safety, tolerability, pharmacokinetics (PK) and early pharmacodynamics (PD) of BGT-002 Tablets.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 and ≤ 65, male or female;
* Body mass index (BMI) ≥ 25 kg/m^2 at screening;
* Subjects fulfilling the following criteria:
* ALT level exceeds the upper limit of normal once within 3 months (ALT elevation without other obvious reasons);
* Mean liver fat content ≥ 10% during screening and at the end of the run-in period (MRI-PDFF);
* Stable body weight (defined as weight gain or loss ≤ 5%) 4-8 weeks pre-dose;
* Pre-dose blood pressure: Systolic blood pressure ≤ 160 mmHg and diastolic blood pressure ≤ 95 mmHg (oral antihypertensive drugs can be taken regularly);
* Maintain the same medication and lifestyle (diet and/or exercise) as those at enrollment during the trial;
* Subjects who have no birth plan from screening to 6 months after the last dose and voluntarily take reliable contraceptive measures;
* Subjects who fully understand the purpose and requirements of the trial, voluntarily participate in the clinical trial, and sign the written ICF, and are able to complete all trial processes according to the trial requirements.

Exclusion Criteria:

* Subjects with a known history of allergies to the test product, any of its components, or related products; as well as those with allergic diseases or an allergic constitution;
* Subjects with heavy alcohol consumption for 3 consecutive months or above within 1 year before screening. "Heavy alcohol consumption" is defined as average daily alcohol consumption of > 20 g for females and > 30 g for males, or uncontrollable alcohol consumption;
* Subjects with cirrhosis suggested by liver biopsy or clinically diagnosed cirrhosis;
* Subjects with other concomitant liver diseases, including but not limited to drug-induced liver disease, alcoholic liver disease, autoimmune liver disease, hemochromatosis, Wilson's disease, suspected or confirmed liver cancer;
* Subjects who have received liver transplantation surgery or plan to have this surgery:
* Subjects who have received bariatric surgery or plan to have this surgery during the study;
* Subjects with type 1 diabetes and poorly controlled type 2 diabetes (HbA1c > 10.5% at screening);
* Patients with diabetes who use hypoglycemic drugs other than metformin;
* Subjects with a history of malignant tumor within 5 years before screening (Note: 1. Subjects with cervical carcinoma in situ whose lesions have been resected and with no evidence of recurrence or metastasis for at least 3 years may participate in this study. 2. Subjects with basal cell or squamous cell carcinoma whose lesions have been completely resected and with no recurrent lesions for at least 3 years can participate in this study;
* Subjects with serious cardiovascular and cerebrovascular events within 6 months before screening, including but not limited to uncontrolled or serious arrhythmia (ventricular fibrillation, atrial fibrillation, etc.), angina unstable, acute myocardial infarction, cardiac failure congestive, coronary intervention (including coronary artery stent implantation, intracoronary thrombectomy, and percutaneous transluminal coronary angioplasty, etc) or coronary artery bypass surgery, peripheral vascular intervention, stroke (except lacunar infarction), and transient ischaemic attack;
* Subjects with gastrointestinal diseases or postoperative conditions affecting drug absorption;
* Subjects who are taking drugs that may cause steatosis/steatohepatitis;
* Subjects who have used ACLY-targeted drugs (Nexletol, etc.) and other study drugs, are taking statins (lovastatin, simvastatin, pravastatin, mevastatin, fluvastatin, atorvastatin, cerivastatin, rosuvastatin, pitavastatin, etc.), fibric acids (such as fenofibrate, gemfibrozil), probucol, warfarin, systemic steroids, cyclosporin or other immunosuppressants, or have taken these drugs less than 1 month or 5 half-lives of the drug (whichever is longer) from the first administration of the study drug;
* Subjects who have used drugs with potential therapeutic effects on NASH (such as GLP-1 receptor agonists, DPP4 inhibitors, SGLT2 inhibitors, or other drugs known to affect liver function and cause steatosis at the discretion of the investigator) during the trial period and within less than 1 month from the screening;
* Subjects with a TG > 6.0 mmol/L, direct bilirubin > 2 × ULN, creatinine clearance < 60 mL/min (calculated using the Cockcroft-Gault formula);
* Platelet count < 75 × 10^9/L;
* Subjects with confirmed positive and clinically significant results for antinuclear antibody (ANA) at screening;
* Subjects with a history of hypothyroidism, hyperthyroidism, or subclinical thyroid disease (except for those with TSH levels < 10 mu/l, normal free T3 and T4 levels, and no symptoms of hypothyroidism);
* Subjects with contraindications to MRI scan;
* Subjects with blood donation or blood loss ≥ 400 mL within 3 months before screening;
* Subjects who have participated in other drug clinical trials within 1 month prior to the screening;
* Pregnant/lactating women or subjects confirmed positive in serum pregnancy test (female);
* Subjects with positive results in urinary drug screening (morphine, marijuana);
* Subjects who have consumed any food or beverage containing alcohol (or positive alcohol breath test result), grapefruit juice/grapefruit juice, methylxanthine (such as coffee, tea, cola, chocolate, and energy drink) within 1 day pre-dose, or have strenuous exercise or other factors affecting drug absorption, distribution, metabolism, and excretion;
* Subjects with other severe systemic diseases unrelated to NASH;
* Subjects infected with viral hepatitis (including hepatitis B and C), AIDS, or syphilis;
* Subjects with high-risk factors of torsades de pointes (hypokalemia, hypomagnesemia, heart rate < 45 bpm), and ECG QTc interval longer than 490 ms during screening;
* Subjects with other factors deemed by investigators as not suitable for the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From Day 1 to Day 56
C-QTc(Concentration-QTc) | Day1、Day28
  To investigate the effect of BGT-002 on QT/QTc interval in subjects

SECONDARY OUTCOMES:
Cmax(Peak Concentration) | Day1
  The peak concentration of BGT-002 tablets was assessed after oral administration of BGT-002
Tmax(Time of maximum observed concentration) | Day1
  Evaluate the time required for the drug to reach its maximum concentration after oral administration of BGT-002
AUC(0-24h)(Area Under Curve) | Day1
  The area under the curve was assessed 0 to 24 hours after oral administration of BGT-002
Cmax,ss | Day28
  The peak concentration at stable state was assessed after oral administration of BGT-002
Tmax,ss | Day28
  The peak time at stable state was assessed after oral administration of BGT-002
AUCss | Day28
  The area under the curve at stable state after the subject's oral administration of BGT-002 was assessed
CLss/F(Steady-State Clearance/bioavailability,F) | Day28
  The clearance rate at stalbe state was assessed after oral administration of BGT-002
Cmin,ss | Day28
  Assess valley concentrations at stable state after oral administration of BGT-002
Rac(Accumulation Ratio) | Day28
  Assess the drug accumulation index after oral administration of BGT-002
MRI-PDFF(Magnetic resonance imaging-derived proton density fat fraction) | Day1 (for subjects with results within 7 days pre-dose, examination may be omitted on Day1), Day29/early withdrawal (+5 days), and Day56 (± 5 days)
  Assess the changes of magnetic resonance imaging derived proton density fat fraction after oral administration of BGT-002
CAP(controlled attenuation parameter) | Day1 (for subjects with results within 7 days pre-dose, examination may be omitted on Day1), Day29/early withdrawal (+5 days), and Day56 (± 5 days)y29、Day56
  Assess the changes of controlled attenuation parameter based on ultrasound after oral administration of BGT-002
LSM(Liver Stiffness Measuremen) | Day1 (for subjects with results within 7 days pre-dose, examination may be omitted on Day1), Day29/early withdrawal (+5 days), and Day56 (± 5 days)
  Assess the changes of liver stiffness measurement after oral administration of BGT-002
BMI(Body Mass Index) | Day1, Day29/early withdrawal, and Day56 (± 5 days)
  Changes of Body Mass Index were assessed after oral administration of BGT-002
ALT(Alanine Aminotransferase) | Day1, Day29/early withdrawal, and Day56 (± 5 days)
  Changes of Alanine Aminotransferase were assessed after oral administration of BGT-002
ASTc(Aspartate Transaminase) | Day1, Day29/early withdrawal, and Day56 (± 5 days)
  Changes of Aspartate Transaminase were assessed after oral administration of BGT-002
TG(Triglyceride) | Day1, Day29/early withdrawal, and Day56 (± 5 days)
  Changes of Triglyceride were assessed after oral administration of BGT-002
LDL-C(Low-Density Lipoprotein Cholesterol) | Day1, Day29/early withdrawal, and Day56 (± 5 days)
  Changes of Low-Density Lipoprotein Cholesterol were assessed after oral administration of BGT-002
TC(total cholesterol) | Day1, Day29/early withdrawal, and Day56 (± 5 days)
  Changes of serum total cholesterol were assessed after oral administration of BGT-002

CONTACTS AND LOCATIONS:
Overall Officials: Ding Yanhua, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT06491576/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT06491576/SAP_001.pdf